CLINICAL TRIAL: NCT04390282
Title: Secondary Prevention and Application-based Lifestyle Support for Patients With Intermittent Claudication
Acronym: PRESIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Christine Kumlien, Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CKtrial2020
Record Dates: First submitted 2020-05-05; First posted 2020-05-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Intermittent Claudication; Vascular Diseases
Keywords: Secondary prevention; Life Style, Healthy; Internet-Based intervention; Illness percetion; Health literacy
MeSH Terms: conditions — Intermittent Claudication; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application-based support system Lifepod®PAD (Experimental): Patients in the experimental group will be introduced to and use Lifepod®PAD, a web-based application designed to support adherence to lifestyle advice and medication for three months. Lifepod®PAD is built as a two-side system. One side is the patient interface, the web-based application, accessible through a smartphone or tablet. The patients can log information about their lifestyle, symptoms and medication and review their data in relation to recommended targets. They get positive feedback, recommendations about healthy behaviours and receive notifications as short messages depending on their individual health status. The other side is the medical interface managed by the health care professionals. All information the patient is reporting into the app can be accessed by the treating nurse and the system ranks the patients, thus gives high priority to patients who have the greatest needs.
  Interventions: Behavioral: Application-based support system
- Life style advice according to usual practice (No Intervention): Patients in the control group will receive usual care meaning advice about lifestyle changes and medication from the physician at the visit in the vascular open clinic.

INTERVENTIONS:
Behavioral: Application-based support system — All participants (experimental and control group) will be invited to a separate appointment at the vascular open clinic at baseline and after three months and measured regarding weight, blood pressure, Ankle Brachial Pressure Index, six minutes walking test and pain. To calculate the estimate 10-year risk of manifesting clinical cardiovascular disease, the Framingham Risk Score will be used. Further, a questionnaire will be answered at baseline and after three months containing the instruments, VascuQoL-6, Health Education Impact Questionnaire and Medication Adherence Report Scale-5.
  Other Names: Life style support according usual clinical practice
  Arms: Application-based support system Lifepod®PAD

SUMMARY:
A randomized controlled pilot trial will be used to test Lifepod®PAD as secondary prevention support system. Approximately 60 patients with intermittent claudication at the Department of vascular diseases at Skåne University hospital will be invited. The intervention group (n=30) will test Lifepod PAD for 3 months and the control group (n=30) will receive secondary prevention as usual. Primary outcome is pain free walking distance and secondary outcomes will be quality of life, illness perception, ankle brachial pressure, self-efficacy, adherence to medical treatment and blood pressure. Acceptability, delivery of the intervention, expected sample size and effect size, procedure of randomization and follow-ups will be evaluated. The outcome will be used to design a main randomized trial. Combinations of quantitative measures and qualitative interviews will be used to understand the process in detail.

DETAILED DESCRIPTION:
A randomized controlled pilot trial will be used to test the application-based support systems Lifepod®PAD that are developed in collaboration with Cross Technology Solutions based on results from our systematic review and previous research testing the Lifepod® system in patients with myocardial infarction.

Sample Approximately 60 patients with intermittent claudication diagnosed at the Department of vascular diseases at Skåne University hospital will be invited to participate. The participants should have access to a smartphone or tablet. For the randomization, envelopes will be prepared by a member of the research group and then mixed by another member of the group. After receiving informed consent, the participants are randomized by drawing one of the sealed envelopes with the information in which group they are included. The trial will have two arms; one group will test Lifepod®PAD (n=30) for three months and one control group (n=30) will receive secondary prevention as usual.

Data collection All participants will be invited to a separate appointment at the vascular open clinic at baseline and after three months and measured regarding weight, blood pressure, ABPI, six minutes walking test and pain. To calculate the estimate 10-year risk of manifesting clinical cardiovascular disease, the Framingham Risk Score will be used. Further, a questionnaire will be answered at baseline and after three months containing the instruments, VascuQoL-6, Health Education Impact Questionnaire (hei-Q) and Medication Adherence Report Scale-5.

Patients randomized to Lifepod®PAD will get access and be introduced to the Lifepod®PAD support system software. Patients in the control group will receive usual care meaning advice about lifestyle changes and medication from the physician at the visit in the vascular open clinic.

After completing the intervention, a random number of patients who have tested Lifepod®PAD will be invited to take part in focus group interviews to discuss their experiences of using the devices. The interviews will be analyzed by thematic content analysis.

The intervention Lifepod®PAD is a web-based application designed to support adherence to lifestyle advice and medication and is built as a two-side system. One side is the patient interface, the web-based application, accessible through a smartphone or tablet. The patients can log information about their lifestyle, symptoms and medication and review their data in relation to recommended targets. They get positive feedback, recommendations about healthy behaviours and receive notifications as short messages depending on their individual health status. The other side is the medical interface managed by the health care professionals. All information the patient is reporting into the app can be accessed by the treating nurse and the system ranks the patients, thus gives high priority to patients who have the greatest needs.

Analysis Primary outcome will be pain free walking distance according to six minutes walking test at baseline and after three months. Secondary outcomes are quality of life, illness perception, self-efficacy, adherence to medical treatment, blood pressure and ABPI. Acceptability, delivery of the intervention, expected sample size and effect size, procedure of randomization and follow-ups will be further evaluated.

Descriptive statistics will be used to describe the study sample. T-tests will be used to compare groups and chi-square tests will be used to study differences in proportions. Effect size will be calculated to estimate the magnitude of the potential effects and constitute a base for power calculation and sample size in a full-size RCT. The outcome will be used to design a main multicenter randomized trial Ethical considerations Verbal and written information about the purpose of the studies will be given and a written informed consent will be obtained in all studies. Additionally, they will be informed that participating is voluntary and the can withdraw at any time without providing any reason. Approval for the project are provided by the Swedish Regional Ethical Review Board (Dnr 2017/609)

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermittent claudication diagnosed at the Department of vascular diseases at Skåne University hospital.

The participants should have access to a smartphone or tablet and be able to speak and understand Swedish.

Exclusion Criteria:

* Patients with intermittent claudication who are considered for revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Pain free walking distance | Change from baseline in pain free walking distance baseline at three months
  Pain free walking distance will be measured by 6 minutes walking test.

SECONDARY OUTCOMES:
Quality of life assessment | Change from baseline in Vascuqol 6 total score (min 6 max 24, higher total score means better quality of life) at three months
  Measured by the quality of life questionnaire Vascuqol 6
Ankle brachial pressure index | Change from baseline in ankle brachial pressure index at three months
  Index based on calculation of ankle pressure and systolic blood pressure
Illness perception | Change from baseline in Illness Perception scale (Include three sections that each have a totalscore, a high totalscore means a personal understanding of illness) at three months
  Measured by Illness Perception Questionnaire
Medication adherence | Change from baseline in Medication Adherence Report Scale (min 5 max 25 in total score a higher total score indicates higher level of adherence) at three months
  Measured by Medication Adherence Report Scale
Self efficacy | Change from baseline in General Self- Efficacy Scale (min 10 max 40 in total score a higher total score indicates more self efficacy) at three months
  Measured by General Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Christine Kumlien, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No